CLINICAL TRIAL: NCT00416208
Title: Consolidation Therapy With Bortezomib in Patients With Multiple Myeloma Aged 61 to 75
Brief Title: Consolidation Therapy With Bortezomib in Elderly Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR006127; 26866138MMY3013 (Other: Janssen-Cilag G.m.b.H, Germany)
Record Dates: First submitted 2006-12-22; First posted 2006-12-27 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Clinical trial; Bortezomib; PS341; Proteasome inhibitor; Consolidation therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bortezomib (Experimental): Bortezomib 1.6 mg/m2 i.v. d1 d8 d15 d22 for 4 cycles each of 35 days
  Interventions: Drug: Bortezomib
- Observation (No Intervention): Observational arm

INTERVENTIONS:
Drug: Bortezomib — 1.6 mg/m2 i.v. d1 d8 d15 d22 for 4 cycles each of 35 days
  Arms: Bortezomib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a consolidation therapy with bortezomib in patients with multiple myeloma aged 61 to 75.

DETAILED DESCRIPTION:
No data supporting the use of bortezomib as a consolidation therapy in multiple myeloma patients are available. Ínterferon tested as consolidation / maintenance therapy has not uniformly proven to prolong survival. In this study the hypothesis is being tested that bortezomib is able to increase duration of response and thus improving survival. This hypothesis is based on the results of the approval study where bortezomib has been tested to improve these endpoints.This is a multicenter, open-label, randomized (patients are assigned to different treatment group by chance) phase III study to evaluate the efficacy and safety of a consolidation therapy with bortezomib in patients with multiple myeloma aged 61 to 75. Three months after receiving high dose melphalan with autologous stem cell transplantation patients will be randomized to receive either consolidation therapy with bortezomib or to be monitored without consolidation therapy. Subjects in the consolidation group will be treated up to 4 cycles (6 weeks each). The main study phase has a duration of 24 weeks. The trial ends after the last enrolled patient has completed a follow-up period of 30 months. The primary objective is to determine the event free survival in treatment and observation group. The secondary objectives are to assess the response rate, overall survival, duration of response, time to progression, short- and long-term toxicities, quality of life and cytogenetic analyses with regard to treatment response, event free survival and overall survival. Primary efficacy analysis: Event free survival is defined as the time from the first disease-related therapeutic procedure until death, progress or relapse. Secondary efficacy analyses: response rate of the treatment group (measured by the relative change of M-protein levels in serum or urine); overall survival is defined as the time from the first therapeutic procedure until death; time to progression is defined as the duration from the date of enrolment until the date of first documented evidence of progressive disease or relapse; duration of response is defined as the duration in months from the date of first evidence of confirmed response to the date of first documented evidence of progressive disease or relapse; quality of life is assessed by the questionnaires EORTC QLQ-C30 (Quality of life questionnaire) and EORTC EQ-5D (Euro Quality of life). Consolidation therapy lasts 4 cycles. Subjects will be treated with bortezomib 1.6 mg/m2 body surface intravenously once weekly for 4 weeks (Days 1, 8, 15, and 22) followed by a 13-day rest period (days 23 to 35). At least 72 hours should relapse between consecutive doses of bortezomib. Therapy should be withheld at the onset of any Grade 3 nonhematological or Grade 4 hematological toxicities excluding neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had pretreatment with single or tandem high dose melphalan therapy and autologous stem cell transplantation as first line therapy
* at least stable disease after stem cell transplantation
* adequate hematological, hepatic and renal lab parameters
* karnofsky status of 70 or more

Exclusion Criteria:

* non-secretory multiple myeloma
* previous treatment with bortezomib
* allogenic stem cell transplantation
* other co-existing malignancy beside basaliome
* peripheral neuropathy
* epilepsia
* other severe comorbidities (renal, hepatic, cardiovascular, metabolic, infectious etc.)
* history of allergic reactions to bortezomib or mannitol
* expected life expectancy of less than 3 months

Ages: 61 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2006-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The difference in event-free survival time will be compared between both arms | Every 35 days during treatment phase, after 4, 8, 12, 18, 24 months during follow-up

SECONDARY OUTCOMES:
Best response to chemotherapy, response rate to chemotherapy , duration of response, toxicities and quality of life; timepoints for assessments will be at end of study, at 1,5 + 4 + 8 +12 + 18 + 24 + 30 months and thereafter 6 monthly | Every 35 days during treatment phase, after 4, 8, 12, 18, 24 months during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H. Clinical Trial, Study Director — Janssen-Cilag G.m.b.H
Locations (37):
- Germany (37):
  - Bamberg
  - Berg
  - Berlin
  - Bremen
  - Dortmund
  - Dresden
  - Duisburg
  - Erlangen
  - Eschweiler
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Goch
  - Göttingen
  - Greifswald
  - Halle
  - Hamburg
  - Hamm
  - Jena
  - Karlsruhe
  - Kempten
  - Kiel
  - Kÿln N/A
  - Lübeck
  - Magdeburg
  - Mutlangen
  - München
  - Münster
  - Nuremberg
  - Oldenburg
  - Regensburg
  - Rostock
  - Stuttgart
  - Trier
  - Ulm
  - Villingen-Schwenningen
  - Wiesbaden
  - Würzburg

REFERENCES:
- [Derived] Straka C, Knop S, Vogel M, Muller J, Kropff M, Metzner B, Langer C, Sayer H, Jung W, Durk HA, Salwender H, Wandt H, Bassermann F, Gramatzki M, Rosler W, Wolf HH, Brugger W, Fischer T, Liebisch P, Engelhardt M, Einsele H. Bortezomib consolidation following autologous transplant in younger and older patients with newly diagnosed multiple myeloma in two phase III trials. Eur J Haematol. 2019 Sep;103(3):255-267. doi: 10.1111/ejh.13281. Epub 2019 Jul 19. PMID 31231828
- [Derived] Einsele H, Knop S, Vogel M, Muller J, Kropff M, Metzner B, Langer C, Sayer H, Jung W, Durk HA, Salwender H, Wandt H, Bassermann F, Gramatzki M, Rosler W, Wolf HH, Brugger W, Engelhardt M, Fischer T, Liebisch P, Straka C. Response-adapted consolidation with bortezomib after ASCT improves progression-free survival in newly diagnosed multiple myeloma. Leukemia. 2017 Jun;31(6):1463-1466. doi: 10.1038/leu.2017.83. Epub 2017 Mar 15. No abstract available. PMID 28293022
- See also: Consolidation therapy with bortezomib in patients with multiple myeloma aged 61 to 75 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=243&filename=CR006127_CSR.pdf